CLINICAL TRIAL: NCT02737189
Title: Randomized Trial of Revascularization With Solitaire Stentriever Versus Best Medical Therapy in the Treatment of Acute Ischemic Stroke Due to Basilar Artery Occlusion Presenting Within 6-24 Hours of Symptom Onset
Brief Title: Basilar Artery Occlusion Chinese Endovascular Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other); The First People's Hospital of Changzhou (Other); Xinqiao Hospital of Chongqing (Other); Changhai Hospital (Other); Baotou Central Hospital (Other); 904th Hospital of the Joint Logistics Support Force of the PLA (Other); Linyi People's Hospital (Other); The 985 Hospital of PLA, Taiyuan, Shanxi (Unknown); The First Affiliated Hospital with Nanjing Medical University (Other); Tianjin TEDA Hospital (Unknown); Liaocheng People's Hospital (Other); Luoyang Central Hospital (Other); Subei People's Hospital of Jiangsu Province (Other); PLA 148 Hospital, Zibo, Shandong (Unknown); Hebei General Hospital (Other); Shengli Oilfield Hospital (Other); Shenzhen Bao'an District People's Hospital (Unknown); The First Hospital of Jilin University (Other); Henan Provincial People's Hospital (Other); Peking University Binhai Hospital (Unknown); Beijing Tiantan Hospital (Other); The Military General Hospital of Beijing, PLA (Unknown); The First Affiliated Hospital of Shanxi Medical University (Other); Beijing Luhe Hospital (Other); Affiliated Hospital of Nantong University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Nanning Second People's Hospital (Other); Chongqing Three Gorges Central Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The Fifth Central Hospital of Tianjin，TianJin (Unknown); Yantaishan Hospital (Unknown); Nanyang Central Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Tianjin Huanhu Hospital (Other); The Affiliated Hospital of Northwest University, Xi'an NO.3 Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Xuanwu201601
Record Dates: First submitted 2016-03-06; First posted 2016-04-13 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2022-05

CONDITIONS: Basilar Artery Occlusion; Ischemic Stroke; Cerebrovascular Disorders
Keywords: Basilar Artery Occlusion; Ischemic Stroke; Mechanical Embolectomy
MeSH Terms: conditions — Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovascular Arm (Experimental): Mechanical embolectomy with Solitaire stentriever in conjunction with manual aspiration
  Best Medical Treatment and maximum supportive care
  Interventions: Procedure: Mechanical embolectomy; Drug: Medical Treatment
- Control Arm (Other): Best Medical Treatment and maximum supportive care, not including mechanical thrombectomy, no intra arterial treatment
  Interventions: Drug: Medical Treatment

INTERVENTIONS:
Procedure: Mechanical embolectomy — Mechanical embolectomy with Solitaire stentriever in conjunction with manual aspiration
  Arms: Endovascular Arm
Drug: Medical Treatment — Best Medical Treatment and maximum supportive care, not including mechanical thrombectomy, no intra arterial treatment

SUMMARY:
Endovascular treatment of acute ischemic stroke has shown strong benefit in several prospective randomized trials in the anterior circulation and endovascular therapy for basilar artery occlusion has shown promising results in several single-arm studies. This has led to a broad adoption of these techniques which are now considered standard of care in many institutions despite the lack of adequate evidence to prove their benefit. Indeed, the rates of symptomatic intracerebral hemorrhage in these studies have consistently been around 5% which raises the question as to whether patients could actually be harmed as opposed to helped by these procedures. This is a prospective, multi-center, randomized, controlled, open, blinded-endpoint trial, with the aim to evaluate the hypothesis that mechanical embolectomy with the Solitaire device is superior to medical management alone in achieving better outcomes in subjects presenting with an acute ischemic stroke caused by occlusion of the basilar artery within 6-24 hours from symptom onset.

DETAILED DESCRIPTION:
Study Objective: To evaluate the hypothesis that mechanical embolectomy with the Solitaire device is superior to medical management alone in achieving favourable outcomes defined as modified Rankin score (mRS) 0-3 at 90 days in subjects presenting with ischemic stroke due to basilar artery occlusion up to 24 hours from symptom onset.

Subject Population: Subjects presenting with acute ischemic stroke within 6-24 hours from symptom onset/last seen well and whose strokes are attributable to an occlusion of the basilar artery. Subjects are either ineligible for IV alteplase or have received IV alteplase therapy without recanalization. The randomization employs a 1:1 ratio of mechanical embolectomy with Solitaire stentriever in conjunction with manual aspiration versus medical management alone. Randomization will be done under a stratification process using age, baseline National Institute of Health Stroke Scale (NIHSS) and therapeutic window. For the primary endpoint, subjects will be followed for 90 days post-randomization.Sample size is projected to be 318 patients.

Care providers: Vascular neurologists and trained interventional neuroradiologists or neurologists in certified comprehensive stroke centers that treat more than 500 acute stroke patients and perform more than 30 acute mechanical thrombectomies every year will treat patients. Neurointerventionalists have to have previously performed at least 10 thrombectomies with Solitaire device in acute ischemic stroke patients.

Interventions: Patients in both arms will be admitted at acute stroke units (or Intensive Care Unit if needed) and treated following the Chinese Guidelines for the Early Management of Patients With Acute Ischemic Stroke. Concomitant medications and non-pharmacological therapies will be recorded. If a decision of stopping support life measures is adopted, this will be recorded in the Case Report Form (CRF).A maximum of six attempts to retrieve the thrombus in a single vessel can be made with any Solitaire device or aspiration. In case an atherosclerotic lesion is found underlying the occlusive lesion angioplasty/stenting through detachment of the Solitaire device will be allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Posterior circulation AIS within 6-24 hours from symptom onset/last seen well where patient is ineligible for i.v. thrombolytic treatment, or patient has received i.v. thrombolytic therapy without recanalization.
2. Occlusion (Thrombolysis in Myocardial Infarction, TIMI 0-1) of the basilar artery or intracranial segments of both vertebral arteries as evidenced by computed tomography (CT) angiography, magnetic resonance (MR) angiography or angiogram.
3. Age ≥18 and ≤80 years.
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score obtained prior to randomization must be equal to or higher than 6 points.
5. No significant pre-stroke functional disability (modified Rankin Scale, mRS ≤ 1).
6. Patient treatable within 24 hours from time last seen well. Isolated vertigo with nausea and/or vomiting is not considered onset of symptom.
7. Informed consent obtained from patient or acceptable patient surrogate.

Exclusion criteria

General Exclusion Criteria:

1. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with international normalized ratio > 3.0.
2. Baseline platelet count < 50.000/µL.
3. Baseline blood glucose < 50mg/dL or > 400mg/dL.
4. Severe, sustained hypertension (systolic blood pressure > 220 mm Hg or diastolic blood pressure > 110 mm Hg).
5. Patients in sedation and/or intubated patients could not be included if baseline NIHSS is not obtained by a neurologist or emergency physician prior to sedation or intubation.
6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS.
7. Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
8. History of life threatening allergy (more than rash) to contrast medium
9. Subjects who has received i.v. tissue plasminogen activator (t-PA) treatment beyond 4.5 hours from the beginning of the symptoms.
10. Patients with acute stroke within the first 48 hours after percutaneous cardiac, cerebrovascular interventions and major surgery (beyond 48h they should be randomized in BAOCHE or excluded for endovascular treatment if poor medical conditions).
11. Renal insufficiency with creatinine ≥ 3 mg/dl.
12. Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
13. Subject participating in a study involving an investigational drug or device that would impact this study.
14. Cerebral vasculitis.
15. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations; mRS score at baseline must be ≤ 1.
16. Unlikely to be available for 90 days follow-up.

Neuroimaging Exclusion Criteria:

1. Hypodensity amounting to a posterior circulation Acute Stroke Prognosis Early CT score (pc-ASPECTS) < 6 and Pons-midbrain-index of ≥ 3 on CT angiography source images or MR with diffusion-weighted imaging or NCCT.
2. CT or MR evidence of hemorrhage (the presence of microbleeds on MRI is allowed).
3. Complete cerebellar infarct on CT or MRI with significant mass effect and compression of the fourth ventricle.
4. Complete unilateral or bilateral thalamic infarction on CT or MRI
5. Evidence of vertebral occlusion, high grade stenosis or arterial dissection in the extracranial or intracranial segment that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment.
6. Subjects with occlusions in both anterior and posterior circulation.
7. Evidence of intracranial tumor (except small meningioma).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2016-07; Primary Completion 2021-09 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients achieving favourable outcomes defined as mRS 0-3 at 90 days | 90 days
  The primary objective of this study is to evaluate the hypothesis that mechanical embolectomy with the Solitaire device is superior to medical management alone in achieving favourable outcomes (mRS ≤ 3) at 90 days in subjects presenting with an acute ischemic stroke caused by occlusion of the basilar artery within 6-24 hours from symptom onset.

SECONDARY OUTCOMES:
Dramatic early favorable response | 24 (-2/+12) hours
  Dramatic early favorable response as determined by an National Institute of Health stroke scale (NIHSS) of 0-2 or NIHSS improvement ≥ 8 points at 24 (-2/+12) hours.
Dichotomized mRS score (0-2 versus 3-6 and 0-4 versus 5-6 ) | 90 days
Proportion of patients achieving meaningful outcomes defined as mRS 0-4 at 12 months. | 12 months
Final infarct volume and the change of infarct volume compared with baseline | 24 hours (-2/+12 hours)
  Infarct volume evaluated on Computed Tomography (CT) or Magnetic Resonance (MR) at 24 hours (-2/+12 hours)
Vessel recanalization with Arterial Occlusive Lesion (AOL) grades | 24 hours (-2/+12 hours)
  Vessel recanalization at 24 hours (-2/+12 hours) in both treatment groups assessed by using Arterial Occlusive Lesion (AOL) grades
Modified Rankin Score (mRS) | 90 days
Barthel Index | 90 days
NIHSS | 90 days
Quality of life analysis | 3 month, 6 months and 1 year
  Quality of life analysis as measured by EuroQol/EQ5D and SF-36 at 3 month, 6 months and 1 year, between interventional therapy vs medical therapy alone
Mortality | at 90 days
Symptomatic intracranial hemorrhage （SICH） | 24 (-2/+12) hours
Serious Adverse Events | 1 year
Montreal Cognition Test (MOCA) | 90 days
Immediate Post-Endovascular Treatment Recanalization (for the Solitaire arm only) | Immediate Post-Endovascular Treatment
  Successful recanalization is defined as TICI (Thrombolysis in Cerebral Infarction) 2b or 3 in the post-procedure angiography.
Procedural related complications | Perioperative period
  arterial perforation, arterial dissection, embolization in a previously uninvolved vascular territory and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, Principal Investigator — Xuanwu Hospital, Beijing; Tudor G Jovin, MD, Principal Investigator — University of Pittsburg Medical Center Stroke
Locations (36):
- China (36):
  - Baotou Central Hospital, Baotou
  - Beijing Luhe Hospital, Beijing
  - Beijing Tiantan Hospital, Beijing
  - The Military General Hospital of Beijing, PLA, Beijing
  - Xuanwu Hospital, Beijing
  - The First People's Hospital of Changzhou, Changzhou
  - Chongqing Three Gorges Central Hospital, Chongqing
  - Xinqiao Hospital of Chongqing, Chongqing
  - Shengli Oilfield Hospital, Dongying
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang
  - First Hospital of Jilin University, Jilin
  - Liaocheng Third People's Hospital, Liaocheng
  - Linyi People's Hospital, Linyi
  - Luoyang Central Hospital, Luoyang
  - Nanjing First People's Hospital, Nanjing
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - Nanning Second People's Hospital, Nanning
  - Nantong University, Nantong
  - Nanyang Central Hospital, Nanyang
  - Changhai Hospital, Shanghai
  - Shenzhen Bao'an District People's Hospital, Shenzhen
  - Hebei General Hospital, Shijiazhuang
  - Second Affiliated Hospital of Soochow University, Suzhou
  - PLA 264 Hospital, Taiyuan
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan
  - Peking University Binhai Hospital, Tianjin
  - The Fifth Central Hospital of Tianjin, Tianjin
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin TEDA Hospital, Tianjin
  - The 101st Hospital of Chinese People's Liberation Army, Wuxi
  - The Affiliated Hospital of Northwest University, Xi'an NO.3 Hospital, Xi'an
  - Subei People's Hospital of Jiangsu Province, Yangzhou
  - Yantaishan Hospital, Yantai
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou
  - Henan Provincial Hospital, Zhengzhou
  - PLA 148 Hospital, Zibo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Zhou M, Wang H, Zhu J, Chen W, Wang L, Liu S, Li Y, Wang L, Liu Y, Yin P, Liu J, Yu S, Tan F, Barber RM, Coates MM, Dicker D, Fraser M, Gonzalez-Medina D, Hamavid H, Hao Y, Hu G, Jiang G, Kan H, Lopez AD, Phillips MR, She J, Vos T, Wan X, Xu G, Yan LL, Yu C, Zhao Y, Zheng Y, Zou X, Naghavi M, Wang Y, Murray CJ, Yang G, Liang X. Cause-specific mortality for 240 causes in China during 1990-2013: a systematic subnational analysis for the Global Burden of Disease Study 2013. Lancet. 2016 Jan 16;387(10015):251-72. doi: 10.1016/S0140-6736(15)00551-6. Epub 2015 Oct 26. PMID 26510778
- [Background] Yang G, Wang Y, Zeng Y, Gao GF, Liang X, Zhou M, Wan X, Yu S, Jiang Y, Naghavi M, Vos T, Wang H, Lopez AD, Murray CJ. Rapid health transition in China, 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Jun 8;381(9882):1987-2015. doi: 10.1016/S0140-6736(13)61097-1. PMID 23746901
- [Background] Liu L, Wang D, Wong KS, Wang Y. Stroke and stroke care in China: huge burden, significant workload, and a national priority. Stroke. 2011 Dec;42(12):3651-4. doi: 10.1161/STROKEAHA.111.635755. Epub 2011 Nov 3. PMID 22052510
- [Background] Lindsberg PJ, Pekkola J, Strbian D, Sairanen T, Mattle HP, Schroth G. Time window for recanalization in basilar artery occlusion: Speculative synthesis. Neurology. 2015 Nov 17;85(20):1806-15. doi: 10.1212/WNL.0000000000002129. PMID 26574535
- [Background] Palaniswami M, Yan B. Mechanical Thrombectomy Is Now the Gold Standard for Acute Ischemic Stroke: Implications for Routine Clinical Practice. Interv Neurol. 2015 Oct;4(1-2):18-29. doi: 10.1159/000438774. Epub 2015 Sep 18. PMID 26600793
- [Background] Powers WJ, Derdeyn CP, Biller J, Coffey CS, Hoh BL, Jauch EC, Johnston KC, Johnston SC, Khalessi AA, Kidwell CS, Meschia JF, Ovbiagele B, Yavagal DR; American Heart Association Stroke Council. 2015 American Heart Association/American Stroke Association Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Oct;46(10):3020-35. doi: 10.1161/STR.0000000000000074. Epub 2015 Jun 29. PMID 26123479
- [Background] Chen CJ, Ding D, Starke RM, Mehndiratta P, Crowley RW, Liu KC, Southerland AM, Worrall BB. Endovascular vs medical management of acute ischemic stroke. Neurology. 2015 Dec 1;85(22):1980-90. doi: 10.1212/WNL.0000000000002176. Epub 2015 Nov 4. PMID 26537058
- [Background] Macleod MR, Davis SM, Mitchell PJ, Gerraty RP, Fitt G, Hankey GJ, Stewart-Wynne EG, Rosen D, McNeil JJ, Bladin CF, Chambers BR, Herkes GK, Young D, Donnan GA. Results of a multicentre, randomised controlled trial of intra-arterial urokinase in the treatment of acute posterior circulation ischaemic stroke. Cerebrovasc Dis. 2005;20(1):12-7. doi: 10.1159/000086121. Epub 2005 May 30. PMID 15925877
- [Background] Yeung JT, Matouk CC, Bulsara KR, Sheth KN. Endovascular revascularization for basilar artery occlusion. Interv Neurol. 2015 Jan;3(1):31-40. doi: 10.1159/000368968. PMID 25999990
- [Background] Punal-Rioboo J, Atienza G, Blanco M. Safety and Efficacy of Mechanical Thrombectomy Using Stent Retrievers in the Endovascular Treatment of Acute Ischaemic Stroke: A Systematic Review. Interv Neurol. 2015 Jul;3(3-4):149-64. doi: 10.1159/000430474. PMID 26279662
- [Background] Akins PT, Amar AP, Pakbaz RS, Fields JD; SWIFT Investigators. Complications of endovascular treatment for acute stroke in the SWIFT trial with solitaire and Merci devices. AJNR Am J Neuroradiol. 2014 Mar;35(3):524-8. doi: 10.3174/ajnr.A3707. Epub 2013 Sep 12. PMID 24029392
- [Background] Hann S, Chalouhi N, Starke R, Gandhe A, Koltz M, Theofanis T, Jabbour P, Gonzalez LF, Rosenwasser R, Tjoumakaris S. Comparison of neurologic and radiographic outcomes with Solitaire versus Merci/Penumbra systems for acute stroke intervention. Biomed Res Int. 2013;2013:715170. doi: 10.1155/2013/715170. Epub 2013 Dec 30. PMID 24490169
- [Background] von Kummer R, Broderick JP, Campbell BC, Demchuk A, Goyal M, Hill MD, Treurniet KM, Majoie CB, Marquering HA, Mazya MV, San Roman L, Saver JL, Strbian D, Whiteley W, Hacke W. The Heidelberg Bleeding Classification: Classification of Bleeding Events After Ischemic Stroke and Reperfusion Therapy. Stroke. 2015 Oct;46(10):2981-6. doi: 10.1161/STROKEAHA.115.010049. Epub 2015 Sep 1. No abstract available. PMID 26330447
- [Background] Wahlgren N, Ahmed N, Davalos A, Ford GA, Grond M, Hacke W, Hennerici MG, Kaste M, Kuelkens S, Larrue V, Lees KR, Roine RO, Soinne L, Toni D, Vanhooren G; SITS-MOST investigators. Thrombolysis with alteplase for acute ischaemic stroke in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST): an observational study. Lancet. 2007 Jan 27;369(9558):275-82. doi: 10.1016/S0140-6736(07)60149-4. PMID 17258667
- [Background] Hacke W, Kaste M, Fieschi C, von Kummer R, Davalos A, Meier D, Larrue V, Bluhmki E, Davis S, Donnan G, Schneider D, Diez-Tejedor E, Trouillas P. Randomised double-blind placebo-controlled trial of thrombolytic therapy with intravenous alteplase in acute ischaemic stroke (ECASS II). Second European-Australasian Acute Stroke Study Investigators. Lancet. 1998 Oct 17;352(9136):1245-51. doi: 10.1016/s0140-6736(98)08020-9. PMID 9788453
- [Background] Puetz V, Sylaja PN, Coutts SB, Hill MD, Dzialowski I, Mueller P, Becker U, Urban G, O'Reilly C, Barber PA, Sharma P, Goyal M, Gahn G, von Kummer R, Demchuk AM. Extent of hypoattenuation on CT angiography source images predicts functional outcome in patients with basilar artery occlusion. Stroke. 2008 Sep;39(9):2485-90. doi: 10.1161/STROKEAHA.107.511162. Epub 2008 Jul 10. PMID 18617663
- [Background] Tomsick T, Broderick J, Carrozella J, Khatri P, Hill M, Palesch Y, Khoury J; Interventional Management of Stroke II Investigators. Revascularization results in the Interventional Management of Stroke II trial. AJNR Am J Neuroradiol. 2008 Mar;29(3):582-7. doi: 10.3174/ajnr.A0843. PMID 18337393
- [Background] Higashida RT, Furlan AJ, Roberts H, Tomsick T, Connors B, Barr J, Dillon W, Warach S, Broderick J, Tilley B, Sacks D; Technology Assessment Committee of the American Society of Interventional and Therapeutic Neuroradiology; Technology Assessment Committee of the Society of Interventional Radiology. Trial design and reporting standards for intra-arterial cerebral thrombolysis for acute ischemic stroke. Stroke. 2003 Aug;34(8):e109-37. doi: 10.1161/01.STR.0000082721.62796.09. Epub 2003 Jul 17. PMID 12869717
- [Background] Liu X, Dai Q, Ye R, Zi W, Liu Y, Wang H, Zhu W, Ma M, Yin Q, Li M, Fan X, Sun W, Han Y, Lv Q, Liu R, Yang D, Shi Z, Zheng D, Deng X, Wan Y, Wang Z, Geng Y, Chen X, Zhou Z, Liao G, Jin P, Liu Y, Liu X, Zhang M, Zhou F, Shi H, Zhang Y, Guo F, Yin C, Niu G, Zhang M, Cai X, Zhu Q, Chen Z, Liang Y, Li B, Lin M, Wang W, Xu H, Fu X, Liu W, Tian X, Gong Z, Shi H, Wang C, Lv P, Tao Z, Zhu L, Yang S, Hu W, Jiang P, Liebeskind DS, Pereira VM, Leung T, Yan B, Davis S, Xu G, Nogueira RG; BEST Trial Investigators. Endovascular treatment versus standard medical treatment for vertebrobasilar artery occlusion (BEST): an open-label, randomised controlled trial. Lancet Neurol. 2020 Feb;19(2):115-122. doi: 10.1016/S1474-4422(19)30395-3. Epub 2019 Dec 9. PMID 31831388
- [Background] Writing Group for the BASILAR Group; Zi W, Qiu Z, Wu D, Li F, Liu H, Liu W, Huang W, Shi Z, Bai Y, Liu Z, Wang L, Yang S, Pu J, Wen C, Wang S, Zhu Q, Chen W, Yin C, Lin M, Qi L, Zhong Y, Wang Z, Wu W, Chen H, Yao X, Xiong F, Zeng G, Zhou Z, Wu Z, Wan Y, Peng H, Li B, Hu X, Wen H, Zhong W, Wang L, Jin P, Guo F, Han J, Fu X, Ai Z, Tian X, Feng X, Sun B, Huang Z, Li W, Zhou P, Tu M, Sun X, Li H, He W, Qiu T, Yuan Z, Yue C, Yang J, Luo W, Gong Z, Shuai J, Nogueira RG, Yang Q. Assessment of Endovascular Treatment for Acute Basilar Artery Occlusion via a Nationwide Prospective Registry. JAMA Neurol. 2020 May 1;77(5):561-573. doi: 10.1001/jamaneurol.2020.0156. PMID 32080711
- [Derived] Jovin TG, Li C, Wu L, Wu C, Chen J, Jiang C, Shi Z, Gao Z, Song C, Chen W, Peng Y, Yao C, Wei M, Li T, Wei L, Xiao G, Yang H, Ren M, Duan J, Liu X, Yang Q, Liu Y, Zhu Q, Shi W, Zhu Q, Li X, Guo Z, Yang Q, Hou C, Zhao W, Ma Q, Zhang Y, Jiao L, Zhang H, Liebeskind DS, Liang H, Jadhav AP, Wen C, Brown S, Zhu L, Ye H, Ribo M, Chang M, Song H, Chen J, Ji X; BAOCHE Investigators. Trial of Thrombectomy 6 to 24 Hours after Stroke Due to Basilar-Artery Occlusion. N Engl J Med. 2022 Oct 13;387(15):1373-1384. doi: 10.1056/NEJMoa2207576. PMID 36239645
- [Derived] Hankey GJ. Endovascular Therapy for Acute Basilar Artery Occlusion. Circulation. 2022 Jul 5;146(1):18-20. doi: 10.1161/CIRCULATIONAHA.122.060571. Epub 2022 Jul 5. No abstract available. PMID 35858168
- [Derived] Li C, Wu C, Wu L, Zhao W, Chen J, Ren M, Yao C, Yan X, Dong C, Song H, Ma Q, Duan J, Zhang Y, Zhang H, Jiao L, Wang Y, Jovin TG, Ji X; BAOCHE Investigators. Basilar Artery Occlusion Chinese Endovascular Trial: Protocol for a prospective randomized controlled study. Int J Stroke. 2022 Jul;17(6):694-697. doi: 10.1177/17474930211040923. Epub 2021 Aug 28. PMID 34427475